CLINICAL TRIAL: NCT01676285
Title: Effect of Metoprolol Succinate in Cardiac Remodeling Related to Nonalcoholic Cirrhosis. Randomized Study.
Brief Title: Metoprolol Succinate in Cardiac Remodeling Related to Cirrhosis
Acronym: CARE Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fernando Bacal, MD; PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0010/11
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Cirrhosis; Cirrhotic Cardiomyopathy; Cardiac Remodeling
Keywords: Cirrhosis; cirrhotic cardiomyopathy; cardiac remodeling; cardiomyopathy; metoprolol succinate; betablockers
MeSH Terms: conditions — Fibrosis; Cardiomyopathies | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metoprolol succinate (Active Comparator): Metoprolol succinate
  Interventions: Drug: Metoprolol succinate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- Follow up (No Intervention): Group without cirrhotic cardiomyopathy, only follow up without randomization.

INTERVENTIONS:
Drug: Metoprolol succinate
  Other Names: Selozok
  Arms: Metoprolol succinate
Drug: placebo
  Arms: Placebo

SUMMARY:
Cirrhotic cardiomyopathy is defined as a chronic cardiac dysfunction in patients with cirrhosis. It is suspected that this specific cardiac dysfunction contributes to the onset of complications in liver disease. The purpose of this prospective, randomized trial is to determine whether metoprolol succinate can revert cardiac dysfunction secondary to cirrhosis (cirrhotic cardiomyopathy), and prevent complications (renal dysfunction, mortality). A total of 100 patients with cirrhotic cardiomyopathy will be randomized (Group R) to receive metoprolol succinate or placebo; other 25 patients without cirrhotic cardiomyopathy (Group F) will only be followed up without medication. All patients will be evaluated in the beginning and again after six months. The assessment protocol includes clinical evaluation, electrocardiogram, echocardiogram, laboratory analysis and life quality questionaire. The end points will be cardiac remodeling, electrophysiologic changes, sympathetic activity, laboratory issue changes, renal function, quality of life, and mortality.

DETAILED DESCRIPTION:
Cirrhotic cardiomyopathy (CMC) is defined as a chronic cardiac dysfunction in patients with cirrhosis. Moreover, it is characterized by an abnormal and blunted response to pathological or pharmacological stress in the absence of any other associated cardiac disease. The diagnostic criteria are: baseline increased cardiac output, attenuated myocardial contractile response to stress, diastolic dysfunction, and electrophysiological repolarization abnormalities. It is suspected that cardiac dysfunction in cirrhosis contribute to the onset of complications in liver disease. We will investigate the effect of metoprolol succinate in the reversal of cardiac dysfunction and prevention of complications of cirrhosis in patients with cirrhotic cardiomyopathy. Furthermore, we want to study the influence of presence of CMC in the evolution of cirrhotic patients. The study will be prospective, randomized, double-blind, and placebo-controlled. The sample consists of 125 patients aged between 18 and 60 years old diagnosed with severe liver cirrhosis (Child B or C or MELD score above 10) with cirrhotic cardiomyopathy or not. Of these, 100 patients with cirrhotic cardiomyopathy will be randomized into two groups: group R1 (metoprolol succinate) and group R2 (placebo). Group F will consist of cirrhotic patients without cardiomyopathy and will not receive medication. Patients will be evaluated by clinical examination, resting electrocardiogram, 24-hour Holter, stress echocardiography and laboratory (brain natriuretic peptide (BNP), catecholamines, plasma renin activity, and troponin) at inclusion and after six months. The end points are: 1) Reversal of cardiac dysfunction in patients with cirrhotic cardiomyopathy, 2) Development of hepatorenal syndrome, 3) Reversal of the electrophysiologic abnormalities, 4)Changes in laboratory tests, and 5) Mortality.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old.
* must have signed the written informed consent.
* nonalcoholic cirrhosis.

Exclusion Criteria:

* Betablockers intolerance;
* Diagnosis of other cardiomyopathy
* Chronicle renal disease (Creatinine > 2.5)
* Heavy alcohol intake history
* Presence of other disease with possible cardiac implication (infiltrative or storage disease)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement of systolic function | six months
  Systolic functional reserve is measured by aortic velocity time integral in echocardiographic at rest and stress with dobutamine.

SECONDARY OUTCOMES:
Improvement in left ventricular diastolic function | six months
Renal function | From randomization until six months
Serum level of BNP, catecholamines, plasmatic renin activity | Six months
Mortality | From randomization until six months of follow up
Quality of life | Six months
Electrophysiologic modifications | Six months
  QT prolongation R-R variability

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bacal, MD, PhD, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- University of Sao Paulo School of Medicine, São Paulo, São Paulo, Brazil